CLINICAL TRIAL: NCT06598176
Title: Developing a Combined Molecular Screening and Triage Test for Cervical Cancer Based on Human Papillomavirus (HPV) Detection, Quantification, Genotyping and DNA Methylation in Self-samples (COMBISCREEN)
Brief Title: Developing a Combined Molecular Screening and Triage Test for Cervical Cancer in Self-samples
Acronym: COMBISCREEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wiebren Tjalma, principal investigator, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B3002023000030
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Uterine Cervical Neoplasm; Uterine Cervical Dysplasia; Human Papilloma Virus; HPV-Related Cervical Carcinoma
Keywords: biomarker; first-void urine; vaginal sample; screening; triage; self-sampling; prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample collection (Experimental): Women will collect one first-void urine sample and one vaginal self-sample at home, one day prior to a scheduled appointment at the hospital. During the hospital visit, an additional clinician collected cervical smear and a blood sample will be collected for the study. In case, the patient also undergoes a surgical intervention for their standard treatment plan, the tissue that is collected there, will also be used and analysed for our study. Cytology and histology results will be used as reference test.
  Interventions: Device: Colli-Pee 20mL device with UCM; Device: Evalyn Brush

INTERVENTIONS:
Device: Colli-Pee 20mL device with UCM — Women will collect a first-void urine (the initial part of the urine stream) sample at home the day before a hospital appointment using the 20mL Colli-Pee device prefilled with urine conservation medium (UCM, Novosanis, Belgium).
Device: Evalyn Brush — Women will collect a vaginal self-sample using the Evalyn Brush (Rovers Medical Devices, The Netherlands) at home the day before a hospital appointment.

SUMMARY:
The goal of the COMBISCREEN project is to develop a fully molecular cervical screening and triage approach that is applicable on self-samples, which are an easily accessible and non-invasive source of biomarkers. The project allows a one-step screening and triage modality and thereby identifies women with clinically relevant disease that are in need of treatment.

DETAILED DESCRIPTION:
Currently, there is still 37% of the Flemish population eligible for cervical cancer screening that remains un(der)screened. Self-collected urine and vaginal samples that can be collected from home and are non-invasive provide an attractive alternative for this group. The aim of this study is to collect different samples from patients with a cervical cancer or a scheduled conization in order to identify potential biomarkers for cervical cancer and cervical intraepithelial neoplasia (CIN). These samples include a home-collected first-void urine (Colli-Pee 20mL prefilled with urine conservation medium (UCM)) and vaginal self-sample (Evalyn Brush), as well as a clinician collected cervical smear, blood sample and when appropriate also a tissue sample. A tissue sample will only be collected when the patient is undergoing surgical procedures for their standard therapy. As such, they do not undergo additional invasive procedures as part of the study. The samples are collected prior to starting therapeutic processes (e.g. conization, chemotherapy, radiotherapy, surgery…). The presence of biomarkers (e.g. human papillomavirus (HPV) and DNA methylation) for cervical cancer and cervical intraepithelial neoplasia (CIN) will be determined and compared in each of the sample types. The results of the biomarker assays will also be compared to clinical results from cytology and histology in order to determine the accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 25 until 64 years old
* Diagnosed with cervical cancer (CIN3+, irrespective of stage) OR in need of conization (irrespective of diagnostic or therapeutic purposes)
* Has not started any form of cancer treatment prior to study enrollment
* Written informed consent must be obtained from patient
* Is able to understand the information brochure and what the study is about

Exclusion Criteria:

* Women that underwent hysterectomy
* Pregnant women or 6 weeks post-partum
* Treatment for cervical (pre)cancer in the last 6 months before participation in the study
* Participating in another interventional clinical study (where e.g., a medical device, drug, or vaccine is evaluated) at the same time of participating in this study. Participation in another observational or low-interventional clinical study at the same time is allowed.
* Unable to give informed consent
* Patient has severe anaemia
* Patient received blood transfusion two weeks before sample collection
* Blood sampling would compromise patients' overall health
* Patients who are positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C.
* Patients who are alcoholic or drug abusers
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, or is not in the best interest of the patient to participate, in the opinion of the investigator.

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2037-02-28 (Estimated)

PRIMARY OUTCOMES:
Detection of (epi)genetic biomarkers for cervical cancer and precancer | 48 months
  A novel assay will be developed for the detection of the human papillomavirus (HPV) and epigenetic biomarkers to determine the presence of cervical (pre)cancer. Using histology outcomes as a reference test.

SECONDARY OUTCOMES:
Comparison of the biomarkers detected in the different sample types. | 48 months
  The biomarkers detected in each of the sample types and their performance will be compared.
Demonstrate non-inferiority of the biomarker assay in self-samples compared to conventional cytology on pap smears. | 48 months
  Demonstrate non-inferiority of the developed biomarker assay in self-samples (index tests) compared to conventional cytology on pap smears (comparator test) for the detection of cervical (pre)cancer, using histology outcomes from tissue samples as reference test.
Determine the predictive value of the biomarker assay and the long-term risk of cervical (pre)cancer | Within 1 year after study completion
  Determine the developed biomarker assay's predictive value and long-term risk of cervical (pre)cancer after an initial test-outcome. Measuring the cumulative incidence of cervical (pre)cancer over time. Using histology outcomes from tissue samples ten years pre- and post-study enrolment as reference test outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Wiebren Tjalma, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universitair Ziekenhuis Antwerpen (UZA), Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No